CLINICAL TRIAL: NCT00257348
Title: A Phase II Trial of Capecitabine and Docetaxel in the Treatment of Advanced and Recurrent Cervical Cancer
Brief Title: Capecitabine and Docetaxel in Advanced/Recurrent Cervical Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Aventis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCI 03-04; 2003-2976 (Other: University of California, Irvine)
Record Dates: First submitted 2005-11-21; First posted 2005-11-22 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2013-02

CONDITIONS: Cervical Cancer
Keywords: Advanced Cervical Carcinoma; Recurrent Cervical Carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Capecitabine; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Capecitabine
Drug: Docetaxel

SUMMARY:
The purpose of the study is to evaluate the effectiveness and side effects of the drugs capecitabine and docetaxel in the treatment of cervical cancer. Capecitabine is approved by the FDA for the treatment of breast and colon cancer. Docetaxel is approved in the treatment of breast and lung cancer. The use of capecitabine and docetaxel in this study for the treatment of cervical cancer is considered investigational. Eligible subjects will take the drug capecitabine (Xeloda) by mouth twice a day every 12 hours, for fourteen consecutive days followed by a 7 day rest period. Subjects will also receive the drug docetaxel (Taxotere) intravenously (in the vein) every three weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically proven stage IVB, recurrent or persistent squamous cell carcinoma, adenosquamous carcinoma, or adenocarcinoma of the cervix which is not amenable to curative treatment with surgery and/or radiation therapy
2. Age greater than or equal to 18
3. All patients must have measurable disease. Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest dimension to be recorded). Each lesion must be greater than or equal to 20 mm when measured by conventional techniques, including palpation, plain x-ray, CT, and MRI, or greater than or equal to 10 mm when measured by spiral CT. Biopsy confirmation is required if the lesion measures < 30 mm or if the treating physician determines it is clinically indicated. Patients must have at least one "target lesion" to be used to assess response on this protocol as defined by Response Evaluation Criteria in Solid Tumors (RECIST). This lesion should be the one that was biopsied if one was performed. Patients with tumors within and outside a previously irradiated field should have the lesion outside of the irradiated area preferentially designated as the "target" lesion.
4. Patients must have adequate:

   * Hematologic function: ANC greater than or equal to 1500/mm3; Platelets greater than or equal to 100,000/mm3; Hemoglobin greater than or equal to 8.0 g/dl
   * Renal function: Serum creatinine less than or equal to 1.2 mg/dl. Patients with a serum creatinine greater than 1.2 mg/dl but less than 1.5 mg/dl must have a 24-hour creatinine clearance determination of > 50 cc/min to be eligible.
   * Hepatic function: Total Bilirubin must be within normal limits. Transaminases (SGOT and/or SGPT) may be up to 2.5 x institutional upper limit of normal (ULN) if alkaline phosphatase is less than or equal to ULN, or alkaline phosphatase may be up to 4 x ULN if transaminases are less than or equal to ULN
5. Patients must have a GOG Performance Status of 0 or 1.
6. Patients must have recovered from the effects of surgery, radiation therapy, or chemoradiotherapy. At least six weeks must have elapsed from the last administration of chemoradiotherapy, and at least three weeks must have elapsed from the last administration of radiation therapy alone.
7. Patients must have signed an approved informed consent form.
8. Patients must be free of clinically active infection.
9. Women of childbearing potential must have a negative pregnancy test. Women of childbearing potential must be willing to consent to using effective contraception while on treatment until they reach menopause.

Exclusion Criteria:

1. Patients with bilateral hydronephrosis which cannot be alleviated by ureteral stents or percutaneous drainage. Patients with a serum creatinine greater than 1.2 mg/dl but less than 1.5 mg/dl with a 24-hour creatinine clearance determination of < 50 cc/min.
2. Patients with a serum creatinine of 1.5 mg/dl or greater.
3. Patients previously treated with chemotherapy except when used concurrently with radiation therapy
4. Patients with a history of severe hypersensitivity reaction to docetaxel, drugs formulated with polysorbate 80, fluoropyrimidine therapy or 5-FU.
5. Patients who are pregnant or lactating
6. Patients with craniospinal metastases or history of craniospinal metastases.
7. Patients with a concomitant malignancy other than non-melanoma skin cancer.
8. Patients with a prior invasive malignancy (except non-melanoma skin cancer) who have had any evidence of disease within the last 5 years or whose prior malignancy treatment contraindicates the current protocol therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2004-03; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Estimate response rate | Weekly
  Complete Response (CR) is disappearance of all target and non-target lesions and no evidence of new lesions documented by two disease assessments at least 4 weeks apart. Normalization of CA125, if elevated at baseline, is required for ovarian carcinoma studies. Partial Response (PR) is at least a 30% decrease in the sum of longest dimensions (LD) of all target measurable lesions taking as reference the baseline sum of LD. There can be no unequivocal progression of non-target lesions and no new lesions. Documentation by two disease assessments at least 4 weeks apart is required.

SECONDARY OUTCOMES:
Determine progression free and overall survival
  Progression free survival-will be calculated from the date of first treatment to the date of disease progression or the date of death or the cut-off date using Kaplan Meier methods.
  Overall survival-will be calculated from the date of first treatment until death or the cut-off date using Kaplan Meier methods.

CONTACTS AND LOCATIONS:
Overall Officials: Bradley J. Monk, MD, Principal Investigator — Chao Family Comprehensive Cancer Center
Locations (1):
- Chao Family Comprehensive Cancer Center, Orange, California, United States